CLINICAL TRIAL: NCT03465085
Title: Streptokinase Versus Unfractionated Heparin Nebulization in Patients With Severe Acute Respiratory Distress Syndrome (ARDS): A Partially Randomized Controlled Trial
Brief Title: Streptokinase Versus Unfractionated Heparin Nebulization in Severe ARDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelaal Ahmed Mahmoud, Associate Professor of Anesthesiology, Beni-Suef University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Heparin-Streptokinase-ARDS
Record Dates: First submitted 2018-03-02; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome
Keywords: ARDS; Streptokinase; Heparin; Nebulization; Inhaled Thrombolytics; Inhaled Anticoagulation
MeSH Terms: conditions — Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — Heparin; Streptokinase

STUDY DESIGN:
Intervention Model Description: Group (I): Heparin group (n=20) received nebulized Heparin 10000 IU/4h. Group (II): Streptokinase group (n=20) received nebulized Streptokinase 250,000 IU/4h.
  Group (III): Control group (n=20) received conservative management
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Investigators prepared and administered the study medication. participants, ICU physician and nurses, and the outcomes assessor were blinded to the two randomized groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Heparin nebulized group (Experimental): Group (I): 20 patients received inhaled Unfractionated Heparin at a dose of 10000 IU/4h by nebulizer, with the total daily dose of nebulized Unfractionated Heparin 60,000 IU
  Interventions: Drug: Unfractionated heparin
- Group II: Streptokinase group (Experimental): Group (II): 20 patients received inhaled Streptokinase at a dose of 250,000 IU/4h by nebulizer, with the total daily dose of nebulized Streptokinase 1,500,000 IU.
  Interventions: Drug: Streptokinase
- Group III: Control group (No Intervention): Twenty patients whom guardian declined to participate actively in the study but accepted to participate passively by consenting for using their data were assigned as Group III or the control group and received conservative management

INTERVENTIONS:
Drug: Unfractionated heparin — Heparin or Streptokinase were nebulized by Aeroneb Pro@ Lab mesh nebulizer (Aerogen Limited, Galway, Ireland) which is incorporated within GE Healthcare's Engström Carestation ventilator (General Electric Company, Finland). Aeroneb nebulizer is a palladium vibrating mesh nebulizer. The central aperture plate of the nebulizer is 5mm in diameter and is perforated with 1000 precision formed holes, that vibrate at 128,000 times per second, to produce the particles with size 1-5 micron in diameter with average MMAD (Mean Mass Aerodynamic Diameter) is 2.1 microns. The nebulized medication (either streptokinase 250,000 IU or heparin 10.000 IU) was prepared in 3 ml volume of distilled water and nebulized for a period of 15 minutes every 4 hours.
  Other Names: Heparin-Sodium Injection 5.000 I.U./ml (B BRAUN)
  Arms: Group I: Heparin nebulized group
Drug: Streptokinase — Heparin or Streptokinase were nebulized by Aeroneb Pro@ Lab mesh nebulizer (Aerogen Limited, Galway, Ireland) which is incorporated within GE Healthcare's Engström Carestation ventilator (General Electric Company, Finland). Aeroneb nebulizer is a palladium vibrating mesh nebulizer. The central aperture plate of the nebulizer is 5mm in diameter and is perforated with 1000 precision formed holes, that vibrate at 128,000 times per second, to produce the particles with size 1-5 micron in diameter with average MMAD (Mean Mass Aerodynamic Diameter) is 2.1 microns. The nebulized medication (either streptokinase 250,000 IU or heparin 10.000 IU) was prepared in 3 ml volume of distilled water and nebulized for a period of 15 minutes every 4 hours.
  Other Names: Streptase (Aventis Behring GmbH, Marburg, Germany U.S)
  Arms: Group II: Streptokinase group

SUMMARY:
Background: Intra-alveolar clotting and alveolar collapse in ARDS is due to alveolar capillaries epithelial and leakage. Subsequently, collapse induces hypoxemia that is resistant to recruitment (RM). Heparin and Streptokinase may prevent or dissolve intra-alveolar fibrin clot respectively helping alveolar re-expansion. We examined and compared the effect of nebulizing Heparin versus Streptokinase on reversing this pathology.

Methods: Sixty severe ARDS (PaO2/FiO2<100) patients and failure of RM, prone position (PP) and neuromuscular block (NMB) were partially randomised into Group (I): (n=20) received nebulized Heparin 10000 IU/4h. Group (II): (n=20) received nebulized Streptokinase 250,000 IU/4h. Group (III): (n=20) received conservative management. Randomization to either Heparin or Streptokinase groups was applied to patients whom guardian accepted participation, while those who declined participation were followed-up as a control. The primary outcome was the change in PaO2/FiO2; the secondary outcomes included the change in compliance, plateau pressure, ventilation-off days, coagulation and ICU mortality.

DETAILED DESCRIPTION:
Methods:

The current study was carried out in the Intensive Care Unit of a tertiary University Hospital following approval by the local Research and Ethics Committee and after obtaining of a written informed consent from the first of kin of the recruited patients.

The guardians of the patients with severe ARDS fulfilling the inclusion criteria of our study were offered to participate in the trial. Randomization to either Heparin or Streptokinase groups was applied to patients whom first of kin agreed to participate in the trial, while patients whom first of kin declined to participate were followed up as a control group. Written informed consent to participate in the trial and to undergo randomization to either Heparin or Streptokinase group was signed by the guardians who approved their patients to participate. Written informed consent to use patients data was signed by the guardians who declined their patients to participate.

Adult patients aged 21-60 years and admitted to our ICU with the diagnosis of ARDS according to Berlin definition (12) were examined and followed up for the presence of the following inclusion criteria;

* Severe ARDS with PO2/FiO2 ratio<100.
* Failure of Recruitment Maneuver (RM), (13) Prone Position (PP) (14) or Neuro-Muscular Block (NMB) (15) to improve hypoxemia.
* No contraindications to thrombolytic or anticoagulant therapy (e.g. Coagulopathy, Heparin-Induced Thrombocytopenia, Previous administration of streptokinase, Known or suspected allergy to heparin or streptokinase, History of intracranial hemorrhage in the past 12 months, Patients with an epidural catheter in place or likely to be placed within the next 48 h.).

Only patients who have all the three criteria were included in the trial following consenting the first of kin.

Sixty severe ARDS patients with failure of RM, PP and NMB and the absence of a contraindication to thrombolytic or anticoagulant therapy were recruited.

Forty patients whom guardian agreed to participate actively in the study were randomly assigned to one of the two groups:

Group (I): 20 patients received inhaled Unfractionated Heparin at a dose of 10000 IU/4h by nebulizer, with the total daily dose of nebulized Unfractionated Heparin 60,000 IU

Group (II): 20 patients received inhaled Streptokinase at a dose of 250,000 IU/4h by nebulizer, with the total daily dose of nebulized Streptokinase 1,500,000 IU.

A random set of numbers were generated by the computer (www.randomizer.org), and each number was sealed in an opaque envelope, and the envelopes were kept in the ICU. One envelope was randomly selected after a patient was selected for recruitment and his/her first of kin consented. The key for assigning numbers to either group was stored on encrypted USB device with one of the investigators. One of the investigators was responsible for preparing the medication nebulizer while the nurse and the ICU physician attending the case and recording the data were blinded to the patients group.

Twenty patients whom guardian declined to participate actively in the study but accepted to participate passively by consenting for using their data, were assigned as Group III, or the control group.

All patients received the routine intensive care protocol for cases of ARDS including the specific ventilatory protocol (16) with monitoring and recording of the following parameters: PaO2 [arterial partial pressure of oxygen], FiO2 [Fraction of inspired oxygen], PaO2/FiO2 ratio, Lung compliance [ml/cmH2o], Peak airway pressure [cmH2o], Coagulation profile [platelets count, prothrombin concentration, INR (International Normalized Ratio), bleeding time] and any side effects or complications as bleeding, coagulopathy, HIT (Heparin Induced Thrombocytopenia) and allergic reactions.

Start and termination of therapy:

Heparin nebulizer or Streptokinase nebulizer (according to the study group) will continue till the occurrence of one or more of the following: (1) Improvement of the hypoxemia as determined by PaO2/FiO2 ratio >300. (2) Improvement of the pulmonary compliance of the patient measured by ventilator defined as dynamic compliance > 50 ml/cmH2O. (3) The occurrence of complications as bleeding or coagulopathy. (4) Failure of the therapy to produce improvement in hypoxemia or compliance after 72 hours of initiation of therapy.

Considering that in case of improvement in either parameter; oxygenation or pulmonary compliance will mandate continuation of therapy for a maximum of 4 days.

Nebulization

Heparin or Streptokinase were nebulized by Aeroneb Pro@ Lab mesh nebulizer (Aerogen Limited, Galway, Ireland) which is incorporated within GE Healthcare's Engström Carestation ventilator (General Electric Company, Finland). Aeroneb nebulizer is a palladium vibrating mesh nebulizer. The central aperture plate of the nebulizer is 5mm in diameter and is perforated with 1000 precision formed holes, that vibrate at 128,000 times per second, to produce the particles with size 1-5 micron in diameter with average MMAD (Mean Mass Aerodynamic Diameter) is 2.1 microns. The nebulized medication (either streptokinase 250,000 IU or heparin 10.000 IU) was prepared in 3 ml volume of distilled water and nebulized for a period of 15 minutes every 4 hours. As per the manufacturer, 0.3 ml of residual volume remains in the nebulizer after each nebulization. Nebulized medications were delivered to the circuit at the junction between the Y-piece and the ETT (Figure 1) to allow the minimal distance between the nebulization delivery port and the ETT. A filter in the expiratory limb (between the ventilator end of the breathing circuit and the ventilator machine) prevented contamination of the circuit. Humidification was supplied by Fisher& Paykel MR 370 humidifier, with the humidifier was stopped and disconnected from the breathing circuit 10 minutes before nebulization and restored 10 minutes after the end of nebulization. During the nebulization, to ensure adequate drug delivery, the ventilatory settings were changed to volume controlled ventilation with TV 500 ml, RR 14/min., I: E ratio of 1:1.5, inspiratory pause 75% of the inspiratory time, PEEP 10 cmH2O with FIO2 of 1. In case of high peak airway pressure ≥40 cmH2O, the tidal volume was decreased gradually to keep peak airway pressure <40 cmH2O. The initial ventilatory settings were restored 10 minutes after the end of nebulization.

The day of start of nebulization is considered day 0 and readings for day 1 was recorded 24 hours after the start of nebulizers.

Ventilation:

A pressure-regulated volume-controlled mode (auto flow) of mechanical ventilation was used. The target tidal volume was set at a range from 4 to 8 ml /kg we started by 6 ml/kg then increased or decreased according to Plateau pressure and CO2 level. Plateau pressure limit up to 30 CmH2o, and CO2 was maintained within normal limit (35 - 45 mmHg), PEEP was maintained 10 mmHg; the Respiratory rate was adjusted according to CO2 level and I: E ratio was maintained at 1: 2. this was routine practice at the time of the study. The trial of weaning used a spontaneous pressure support mode. The level of pressure support was adjusted to maintain the target tidal volume. Extubation was considered if patients meet the criteria of weaning such as being hemodynamically stable and cooperative in addition to minimal ventilator parameter (SpO2> 95% on a pressure support mode < 10 cm H2O, PEEP < 5 cm H2O and FiO2 < 50%).

Outcomes

The primary outcome was the mean daily ratio of PaO2 to FiO2 (PaO2/FiO2). The Secondary outcomes included; static lung compliance, plateau pressure, change in PaCO2, ventilator-off days in surviving patients at ICU discharge, ICU mortality at discharge from ICU and coagulation profile and occurrence of any bleeding complications.

Sample size estimation and Statistical analysis:

Sample size calculated after obtaining preliminary data from 5 patients in control group that revealed mean (SD) of PaO2/FiO2 ratio at day 8 was 82(13). Assuming 30% difference between groups and by using G power software (version 3.1.3, Düsseldorf, Germany) with power 95% and alpha error and with doubling SD, total sample size was 57 patients rolled up to 60 for possible dropout.

The data were examined for normality of distribution by Kolmogorov-Smirnov test (P <0.05). Continuous variables with normal distribution were expressed as mean ± SD (range) and were compared for significant differences between groups by using independent t-test. Paired t-test was used for intragroup comparisons between day-1 and day-8 for each group. Comparison of the means of normally distributed data was done using Two-way analysis (Two Factors (Group and Time)) of variance (between within mixed design) to test Group, Time and Group*Time interaction. The categorical variables were presented in numbers and were compared for significance by using chi squared (χ2) test or Fisher's exact test when appropriate. For all comparisons, a P value < 0.05 will be considered significant. IBM SPSS Advanced Statistics Version 22.0 was used for Data Analysis (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Severe ARDS with PO2/FiO2 ratio<100.
* Failure of Recruitment Maneuver (RM), Prone Position (PP) or Neuro-Muscular Block (NMB) to improve hypoxemia.
* No contraindications to thrombolytic or anticoagulant therapy (e.g. Coagulopathy, Heparin-Induced Thrombocytopenia, Previous administration of streptokinase, Known or suspected allergy to heparin or streptokinase, History of intracranial hemorrhage in the past 12 months, Patients with an epidural catheter in place or likely to be placed within the next 48 h.).
* Static compliance <50 ml/cmH2O

Exclusion Criteria:

* PO2/FiO2 ratio>100.
* The success of Recruitment Maneuver (RM), Prone Position (PP) or Neuro-Muscular Block (NMB) to improve hypoxemia.
* Contraindications to thrombolytic or anticoagulant therapy (e.g. Coagulopathy, Heparin-Induced Thrombocytopenia, Previous administration of streptokinase, Known or suspected allergy to heparin or streptokinase, History of intracranial hemorrhage in the past 12 months, Patients with an epidural catheter in place or likely to be placed within the next 48 h.)
* Static compliance >50 ml/cmH2O

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Change in PaO2/FiO2 ratio | daily over eight days
  Change in the ratio of arterial oxygen tension to fraction of inspired oxygen from the baseline (day 0, before randomization and or the start of intervention) to day 1 to day 8 after the randomization and or start of intervention.

SECONDARY OUTCOMES:
Change in the plateau pressure | daily over eight days
  Change in the plateau airway pressure during ventilation from the baseline (day 0, before randomization and or the start of intervention) to day 1 to day 8 after the randomization and or start of intervention.
Change in the pulmonary compliance | daily over eight days
  change in volume of the lungs per change in pressure during ventilation from the baseline (day 0, before randomization and or the start of intervention) to day 1 to day 8 after the randomization and or start of intervention.
ICU survival rate | At the end of ICU stay up to one year after the start of recruitment
  Number of patients who are discharged alive
ICU length of stay | At the end of ICU stay up to one year after the start of recruitment
  the total duration the patient stays in ICU
Tracheostomy rate | During ICU stay up to one month after the start of recruitment
  number of patients who required tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Hatem Elmoutaz Mahmoud, MD, Study Director — Beni-Suef University

IPD SHARING:
Plan to Share IPD: Undecided